CLINICAL TRIAL: NCT00975988
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance (PMS) to Monitor the Safety and Effectiveness of TYKERB® Tablets Administered in Korean Patients According to the Prescribing Information
Brief Title: Regulatory TYKERB® Tablets PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112477
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Cancer
Keywords: PMS (post-marketing surveillance); TYKERB® tablets
MeSH Terms: conditions — Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TYKERB® tablets: There is only one group. This group includes patients administrated TYKERB® tablets
  Interventions: Drug: TYKERB® tablets

INTERVENTIONS:
Drug: TYKERB® tablets — Patients administrated TYKERB® tablets according to the prescribing information

SUMMARY:
Non-interventional, open-label, single group, multicentric post-marketing surveillance to monitor the safety and effectiveness of TYKERB® tablets administered in Korean patients according to the prescribing information TYKERB® is a registered trademark of the GlaxoSmithKline group of companies.

DETAILED DESCRIPTION:
Non-interventional, open-label, single group, multicentric post-marketing surveillance to monitor the safety and effectiveness of TYKERB® tablets administered in Korean patients according to the prescribing information

TYKERB® tablets will be administered with capecitabine for HER2 overexpressing advanced or metastatic breast cancer treatment or with letrozole for the treatment of postmenopausal women with hormone receptor positive metastatic breast cancer that overexpresses the HER2 as described the prescribing information of TYKERB® tablets

ELIGIBILITY:
All subjects must satisfy the following criteria at PMS entry according to MFDS PMS regulation:

* Subjects with indication in the locally approved prescribing information
* Subjects with no contraindication according to the prescribing information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated TYKERB® tablets at the site
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events after TYKERB® tablets administration | 12 months

SECONDARY OUTCOMES:
Effectiveness of TYKERB® tablets and Occurrence of unexpected adverse drug reaction and serious adverse event after TYKERB® tablets administration | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea